CLINICAL TRIAL: NCT00003536
Title: Phase II Randomized Study of Methotrexate With or Without Antineoplaston A10 Capsules in Women With Advanced Breast Cancer
Brief Title: Methotrexate With or Without Antineoplaston Therapy in Treating Postmenopausal Women With Advanced Refractory Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BC-BR-10; CDR0000066584 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-12

CONDITIONS: Stage IV Breast Cancer; Recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — antineoplaston A10; Methotrexate; Biological Therapy; Drug Therapy; Complementary Therapies

INTERVENTIONS:
Drug: antineoplaston A10
Drug: methotrexate
Procedure: alternative product therapy
Procedure: biological therapy
Procedure: biologically based therapies
Procedure: cancer prevention intervention
Procedure: chemotherapy
Procedure: complementary and alternative therapy
Procedure: differentiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Antineoplastons are naturally occurring substances that may also be made in the laboratory. Antineoplastons may inhibit the growth of cancer cells. It is not yet known whether giving antineoplastons with chemotherapy is more effective than chemotherapy alone in treating women with refractory breast cancer.

PURPOSE: This randomized phase II trial is studying methotrexate alone to see how well it works campared to methotrexate and antineoplaston therapy in treating postmenopausal women with advanced refractory breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the antitumor activity of antineoplaston A10 with methotrexate vs methotrexate alone, in terms of objective tumor response, in women with advanced breast cancer.
* Compare the adverse effects of and tolerance to these regimens in these patients.

OUTLINE: This is a randomized study.

* Arm I: Patients receive gradually escalating doses of oral antineoplaston A10 capsules 7 times daily until the maximum tolerated dose is reached, followed by oral methotrexate capsules 2 to 3 times per day in five days on and five days off courses. Treatment continues in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral methotrexate alone on the same schedule as in arm I.

Tumors are measured every 4 months for 2 years, every 6 months for years 3 and 4, and then annually for years 5 and 6.

PROJECTED ACCRUAL: A total of 30-70 patients will be accrued for this study within at least 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced breast cancer that is refractory or unlikely to respond to hormonal therapy AND failed at least 1 prior chemotherapy regimen
* Symptomatic lymphangitic pulmonary dissemination allowed
* Extensive visceral metastasis allowed
* Patients who are refractory or who have failed to respond after at least 8 weeks of methotrexate or a methotrexate-containing regimen are not eligible
* Measurable disease
* No bone metastases
* Hormone receptor status:
* Estrogen receptor negative

PATIENT CHARACTERISTICS:

Age:

* Postmenopausal

Sex:

* Female

Menopausal status:

* Postmenopausal

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT no greater than 2 times normal
* Blood ammonia normal
* No hepatic failure

Renal:

* BUN less than 60 mg/dL
* Creatinine no greater than 2.5 mg/dL
* Creatinine clearance greater than 60 mL/min
* No chronic renal failure

Cardiovascular:

* No severe heart disease

Pulmonary:

* No severe lung disease

Other:

* No serious active infections or fever
* No other concurrent serious disease
* No prior or concurrent secondary malignancies within the past 2 years
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent biologic therapy for metastatic breast cancer

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior cytotoxic chemotherapy and recovered
* No other concurrent chemotherapy for metastatic breast cancer

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior hormonal therapy and recovered
* No concurrent hormonal therapy for metastatic breast cancer

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy for metastatic breast cancer

Surgery:

* Not specified

Other:

* At least 4 weeks since prior participation in experimental clinical trials
* No prior antineoplaston A10 therapy
* No other concurrent treatment for metastatic breast cancer
* No concurrent salicylates, nonsteroidal anti-inflammatory drugs, phenylbutazone, phenytoin, and sulfonamides

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Study Chair — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States